CLINICAL TRIAL: NCT03434678
Title: Randomized Controlled Trial of Epidural-General Anesthesia Versus General Anesthesia for Open Pancreaticoduodenectomy: Influence on Complications and Overall Two Year Survival
Brief Title: Use of Epidurals Intraoperatively for Patients Undergoing Pancreas Resection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18-056
Record Dates: First submitted 2018-02-08; First posted 2018-02-15 (Actual); Results first posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2024-07

CONDITIONS: Pancreatic Cancer
Keywords: General Anesthesia; Epidural; Pancreaticoduodenectomy; 18-056
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Bupivacaine; Fentanyl

STUDY DESIGN:
Intervention Model Description: Prospective randomized controlled single institution trial.
Who Masked: Investigator
Masking Description: (surgical staff) blinded
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Epidural-General Anesthesia (Experimental)
  Interventions: Drug: Propofol+ Rocuronium+ Fentanyl 2 mcg/kg+ Inhalational Agent, Bupivacaine 0.125% + Fentanyl 5 mcg/ml; Procedure: Open Pancreaticoduodenectomy
- General Anesthesia (Active Comparator)
  Interventions: Drug: Propofol+ Rocuronium+ Fentanyl + Inhalational; Procedure: Open Pancreaticoduodenectomy

INTERVENTIONS:
Drug: Propofol+ Rocuronium+ Fentanyl 2 mcg/kg+ Inhalational Agent, Bupivacaine 0.125% + Fentanyl 5 mcg/ml — Patient will have their epidural started at the beginning of the surgery and receive fewer opioid drugs. The epidural is continued into the recovery room.
  Arms: Epidural-General Anesthesia
Drug: Propofol+ Rocuronium+ Fentanyl + Inhalational — Patient will have the standard intraoperative management during surgery and have the epidural started just before being taken to the recovery room.
  Arms: General Anesthesia
Procedure: Open Pancreaticoduodenectomy — Whipple' Procedure

SUMMARY:
The purpose of this study is to see if there is a difference in complications in patients who have an epidural started earlier (during their surgery) and used as part of the anesthetic in addition to using it for post operative pain compared with patients who receive an epidural later in the surgery to be used only for post operative pain.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥ 18 years of age who can provide informed consent
* Scheduled for pancreaticoduodenectomy

Exclusion Criteria:

* Pregnancy
* History of documented anaphylaxis or contraindication to any of the study medications
* Significant cognitive impairment or documented psychologic impairment
* Contraindication to epidural per Pain Service guidelines
* Use of a sustained release opioid medication such as long-acting morphine, fentanyl patches, methadone, and buprenorphine within the last 3 months
* Post randomization exclusion will occur if the patient is found to have unresectable disease at laparotomy and therefore will not have the potential for the same postoperative complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2018-01-30 (Actual); Primary Completion 2024-07-10 (Actual); Study Completion 2024-07-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Florence Grant, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (3):
- United States (3):
  - Memorial Sloan Kettering Basking Ridge (Consent only), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Commack (Consent only), Commack, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Epidural-General Anesthesia | General Anesthesia
Started | 65 | 68
Completed | 50 | 54
Not Completed | 15 | 14
Not completed — Withdrawal by Subject | 13 | 13
Not completed — Found to be ineligible post randomization | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Epidural-General Anesthesia | General Anesthesia | Total
Number analyzed (Participants) | 50 | 54 | 104
Age, Continuous [Median (Full Range); unit: years] | 66 [44 to 82] | 68 [41 to 85] | 67 [41 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 25 | 40
  Male | 35 | 29 | 64
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 2 | 7
  Not Hispanic or Latino | 42 | 47 | 89
  Unknown or Not Reported | 3 | 5 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 4 | 5
  Native Hawaiian or Other Pacific Islander | 4 | 0 | 4
  Black or African American | 4 | 4 | 8
  White | 41 | 45 | 86
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 50 | 54 | 104

OUTCOME MEASURES:

1. Primary Outcome: Number of Incidences of Grade 3 or Greater Complications
Description: Complications will be graded in severity according to the MSKCC Graded Post Operative Complications Criteria based on the modified Dindo, Clavien classification of surgical complications, a grading system commonly used for this procedure.3,4 This classification grades complications from 1-5, with Grade 1 complications requiring bedside intervention. Grade 2 requires moderate interventions, such as intravenous medications. Grade 3 requires either a surgical, endoscopic or interventional radiology procedure for treatment. Grade 4 results in chronic deficit or disability. Grade 5 complications result in death.
Time Frame: 90 days post operatively
Measure: Number; unit: Number of complications
Arm/Group | Epidural-General Anesthesia | General Anesthesia
Number analyzed (Participants) | 50 | 54
Number of complications | 0 | 0

ADVERSE EVENTS:
Time Frame: 90 days post operatively
Arm/Group | Epidural-General Anesthesia | General Anesthesia
All-Cause Mortality (participants affected / at risk) | 23/50 | 24/54
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/54
Other Adverse Events (participants affected / at risk) | 0/50 | 0/54

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-02): https://cdn.clinicaltrials.gov/large-docs/78/NCT03434678/Prot_SAP_001.pdf